CLINICAL TRIAL: NCT01913782
Title: The Impact of Epidural Steroid Analgesia on Functional MRI for Patients With Low Back Pain
Brief Title: The Impact of Epidural Steroid Analgesia on Functional MRI for Patients With LBP
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Yen Chin Liu, Visiting Staff, Department of Anesthesiology Chief, National Cheng-Kung University Hospital
Other Study IDs: B-ER-101-143
Record Dates: First submitted 2013-07-25; First posted 2013-08-01 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic low back pain, CLBC, fMRI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — fMRI image
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients with low back pain: 1. Patients with disc herniation or radiculitis who are over 18 years of age.
  2. Patients with a history of chronic function-limiting low back pain and lower extremity pain for at least one months' duration.
  3. Patients who are competent to understand the study and provide written informed consent and participate in outcome measurements.

SUMMARY:
Chronic low back pain (CLBP) is the most prevalent form of chronic pain, and the most common reason for disability in working-age population [2]. CLBP has also been reported associated with many abnormal brain anatomy and function which includes the reduction in cortical gray matter in the bilateral dorsolateral prefrontal cortex (DLPFC), thalamus, brain stem, primary somatosensory cortex, and posterior parietal cortex. [3-5] There are already many studies that demonstrated abnormal cortical function for people with CLBP [6-10]. Meanwhile, DLPFC was also reported to be influenced by many pain process which included pain modulation [11-13], placebo analgesia [14, 15], pain control [16, 17]or pain catastrophizing[18]. And recent report has showed that effective treatment of chronic back pain patients reverses abnormal DLPFC function[19]. Meanwhile, epidural steroid injection has been performed in clinical for routinely managed for low back pain patients. Patients refused or have no indication for surgery or have little response to rehabilitation may consider this management. There was good evidence for short- and long-term relief of chronic pain secondary to disc herniation with local anesthetic and steroids[20, 21]. However, the impact of this treatment on functionalMRI (fMRI) has never been investigated. The investigators research will try to solve this issue.

This study will provide a good relationship for the pain fMRI image in brain after local lumbar spine management. And the investigators also want to perform the first data that showed local lumbar analgesia have the impact on brain image change.

DETAILED DESCRIPTION:
Pain, as an ancient enemy to human kind, was one of the most mystical phenomena within our body. For centuries, people search the magic wand to solve this issue and reach the heaven destination. However, like our original sin commit by Adam and Eve, the shadow of pain always surround and even rebel our body and spirit. Even more, pain traps our soul and body not only for the acute stage induced by noxious stimulation but also change our mind and body whenever chronic period start even the stimulation disappears. Chronic pain so far has become one of the greatest health issues for modern people. Chronic pain affects millions of people and the treatment options are quite limited and not effective everyone[1]. On the other way, why and how people develop chronic pain, especially when there is no further painful stimulation, remain to be investigated.

Chronic low back pain (CLBP) is the most prevalent form of chronic pain, and the most common reason for disability in working-age population [2]. CLBP has also been reported associated with many abnormal brain anatomy and function which includes the reduction in cortical gray matter in the bilateral dorsolateral prefrontal cortex (DLPFC), thalamus, brain stem, primary somatosensory cortex, and posterior parietal cortex. [3-5] There are already many studies that demonstrated abnormal cortical function for people with CLBP [6-10]. Meanwhile, DLPFC was also reported to be influenced by many pain process which included pain modulation [11-13], placebo analgesia [14, 15], pain control [16, 17]or pain catastrophizing[18]. And recent report has showed that effective treatment of chronic back pain patients reverses abnormal DLPFC function[19]. Meanwhile, epidural steroid injection has been performed in clinical for routinely managed for low back pain patients. Patients refused or have no indication for surgery or have little response to rehabilitation may consider this management. There was good evidence for short- and long-term relief of chronic pain secondary to disc herniation with local anesthetic and steroids[20, 21]. However, the impact of this treatment on functionalMRI (fMRI) has never been investigated. The investigators research will try to solve this issue.

Patients who first visited in pain clinic for low back pain with root sign will be included in this study.

Inclusion Criteria: 1. Patients with disc herniation or radiculitis who are over 18 years of age. 2. Patients with a history of chronic function-limiting low back pain and lower extremity pain for at least one months' duration. 3. Patients who are competent to understand the study and provide written informed consent and participate in outcome measurements. Exclusion Criteria: Patients have previous lumbar surgery with metal instrument. Initial MRI shows spinal stenosis or without disc herniation. Patients have unstable opioid use, uncontrolled psychiatric disorders, uncontrolled acute medical illness, any condition that could interfere with the interpretation of outcome assessments, pregnant or lactating women or allergy to local anesthetics or steroid. Patients who are unable to perform MRI or fMRI will also be excluded.

Pre-enrollment evaluation included demographic data, medical and surgical history with coexisting disease, lumbar spine X-ray will also be performed.

After physical neurological examinations, pain questionnaire will be applied for initial pain evaluation which includes pain intensity and character and physical activity and emotion influence form their pain. Patients then will be performed the first MRI/fMRI study (with the MRI informed consent, appendix B) for their lumbar spine and brain condition. Anyone who don't have shown spine problem will be excluded for epidural steroid injection. After patients' MRI/fMRI evaluation, caudal epidural steroid injection (Regiment: 0.2% lidocaine plus kenacort 40 mg for 20 ml,) will then be performed in pain therapy room ( with the Epidural informed consent, appendix C). Caudal epidural block will be performed 2-3 times with 2 week interval to reach optimal analgesia. The pain condition will be followed every month with pain questionnaire for up 3 month. The secondary MRI/fMRI will then be performed 3 months later after the first caudal epidural steroid injection.

MRI scans will be acquired on a 3T scanner in NCKU. The special technician will help us and the patient for MRI scan and the setting of all MRI parameter. Dr. Sun and a qualified radiologist will help for data analysis after MRI performance. The investigators will also follow the method that described before[19]: An anatomical scan will be acquired at the beginning of the session and lasted 5 min. The following parameters will be used: echo time (TE) 3 ms, repetition time (TR) 2.3 s, flip angle 9。, resolution 1*1*1 mm. During a functional scan of ~5 min, subjects will perform the Multi-Source Interference Task as previous reported[22, 23]. The task stimuli will be presented on a screen in the subjects' view while lying in the MRI scanner, and subjects will respond on a three-button response box. The task has three levels of difficulty, a motor control task, and easy level and a difficult level. The task will enhance the brain network if pain persistent[23]. The parameters for functional scan were as follow: echo-planar imaging, TE 3 ms, TR 2.26s, flip angle 90。, 128 frames, 64*64 matrix, 38 slices for whole-brain coverage, resolution 4*4*4 mm. Images were acquired in the axial plane, plus 30。 from the anterior commissure-posterior commissure line to avoid the eyes. The fMRI data analysis will be help under our university team.

Total patients number will be calculated on the basis of significant pain relief and set as 33 patients with the following statistic parameter: α: 0.05(type I error probability), power 0.8(probability of correctly rejecting the null hypothesis), δ:0.5(difference in population means), σ:1(standard deviation of difference). 20 % noncompliance rate was added and total 40 patients will be included in this study. According to previous report, 20 more low back patients (oral pain control drug plus rehab and refuse epidural steroid injection) were needed to include for twice MRI survey.[19]

Statistical analysis will include the chi-square, Fisher exact test, t test and paired t test. The chi-square will be used to test the difference in proportions. Fisher exact test will be for whatever the expected value is less than 5; paired t test will used for comparing the pre-and post-treatment results. For comparison of mean between groups, t test will be done. All the data will be presented as mean ± SEM, and P < 0.05 will be considered statistically significant in all cases.

This study will provide a good relationship for the pain fMRI image in brain after local lumbar spine management. And the investigators also want to perform the first data that showed local lumbar analgesia have the impact on brain image change.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with disc herniation or radiculitis who are over 18 years of age.
2. Patients with a history of chronic function-limiting low back pain and lower extremity pain for at least one months' duration.
3. Patients who are competent to understand the study and provide written informed consent and participate in outcome measurements.

Exclusion Criteria:

* Patients have previous lumbar surgery with metal instrument. Initial MRI shows spinal stenosis or without disc herniation. Patients have unstable opioid use, uncontrolled psychiatric disorders, uncontrolled acute medical illness, any condition that could interfere with the interpretation of outcome assessments, pregnant or lactating women or allergy to local anesthetics or steroid. Patients who are unable to perform MRI or fMRI will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who first visited in our pain clinic for low back pain with root sign will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
The pain fMRI image in brain after local lumbar spine | 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Chin Liu, Doctor, Study Chair — Department of Anesthesiology, National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Shengli Rd, Taiwan